CLINICAL TRIAL: NCT01140464
Title: Adolescent Collaborative Care Treatment for Depression
Brief Title: Reaching Out to Adolescents With Depression
Acronym: ROAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Kaiser Permanente (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Laura Richardson, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01MH085645 (NIH); R01MH085645 (NIH)
Record Dates: First submitted 2010-06-01; First posted 2010-06-09 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Depression
Keywords: Adolescents
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Usual Care (Active Comparator): Usual care treatment of depression in primary care settings. Usual care considered enhanced as patients and their parents were given screening results and encouraged to seek care from their primary care doctor and behavioral health services.
  Interventions: Other: Enhanced Usual Care
- Collaborative Care (Active Comparator): Collaborative care intervention for depression. Involves care management, evidence based treatments in primary care setting, symptom monitoring and stepped care design
  Interventions: Other: Collaborative care

INTERVENTIONS:
Other: Collaborative care — Provision of depression care management in the primary care setting to improve delivery of evidence based treatments
  Arms: Collaborative Care
Other: Enhanced Usual Care — Provision of screening results to provider, teen and parent with recommendation to seek further care
  Arms: Enhanced Usual Care

SUMMARY:
Major Depression is one of the most common mental health disorders in adolescence and is associated with significant impairments in development and functioning. This project will rigorously test the Adolescent Collaborative Care Treatment intervention, a health services intervention designed to improve management for depressive disorders among adolescents, via a randomized controlled trial comparing the intervention to usual care. Key components of the trial include enhanced education for youth and parents, youth involvement in choice of evidence-based treatments, care management by an allied health professional with regular supervision by a mental health specialist and pediatrician, and stepped care to advance treatment when youth are not improving. Additional features have been added to engage adolescents and parents including a moderated message board for youth to share with and learn from one another, formalized involvement of the parent, and availability of the care manager during after school hours. Our findings will provide key information on the effectiveness of a developmentally-sensitive adapted collaborative care intervention for the treatment of adolescent depression.

ELIGIBILITY:
Inclusion Criteria:

* depression
* age 13-17 years
* enrollment in study Primary Care Clinics

Exclusion Criteria:

* suicidality
* already enrolled Specialty mental health care
* mental health hospitalization in the prior year
* substance abuse
* bipolar disorder
* non-English speaker

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2010-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Child Depression Rating Scale | 12 months
  Depressive symptoms

SECONDARY OUTCOMES:
Columbia Impairment Scale | 12 months
  Functional impairment

CONTACTS AND LOCATIONS:
Locations (1):
- Group Health Cooperative, Seattle, Washington, United States

REFERENCES:
- [Derived] Wright DR, Haaland WL, Ludman E, McCauley E, Lindenbaum J, Richardson LP. The Costs and Cost-effectiveness of Collaborative Care for Adolescents With Depression in Primary Care Settings: A Randomized Clinical Trial. JAMA Pediatr. 2016 Nov 1;170(11):1048-1054. doi: 10.1001/jamapediatrics.2016.1721. PMID 27654449
- [Derived] Richardson LP, Ludman E, McCauley E, Lindenbaum J, Larison C, Zhou C, Clarke G, Brent D, Katon W. Collaborative care for adolescents with depression in primary care: a randomized clinical trial. JAMA. 2014 Aug 27;312(8):809-16. doi: 10.1001/jama.2014.9259. PMID 25157724